CLINICAL TRIAL: NCT00386607
Title: A 54-week, Open-label, Multicenter Study to Assess the Long-term Safety and Tolerability of the Combination of Aliskiren 300 mg /Valsartan 320 mg in Patients With Essential Hypertension Followed by a 26 Week Open-label Extension to Assess the Long-term Safety and Tolerability of the Triple Combination of Aliskiren/Valsartan/Hydrochlorothiazide(HCTZ)
Brief Title: A Safety and Tolerability Study of the Combination of Aliskiren/Valsartan in Patients With High Blood Pressure, Followed by Long-term Safety and Tolerability of Aliskiren, Valsartan and Hydrochlorothiazide.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPV100A2301; CSPV100A2301E1
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, valsartan, HCTZ, blood pressure
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Valsartan; Hydrochlorothiazide

ARMS (2):
- Core Treatment (Experimental): Oral pills of aliskiren 150 mg /valsartan 160 mg in combination for 2-weeks. The aliskiren 300 mg /valsartan 320 mg in combination for 52-weeks, optional addition of Hydrochlorothiazide (HCTZ) 12.5 mg starting from Week 10 if the blood pressure was uncontrolled (mean sitting Systolic Blood Pressure ≥ 140 and/or mean sitting Diastolic Blood Pressure ≥ 90 mmHg). The dose of Hydrochlorothiazide (HCTZ) 12.5 mg could be increased to 25 mg if blood pressure remained uncontrolled.
  Interventions: Drug: Aliskiren; Drug: Valsartan
- Extension Treatment (Experimental): For patients entering into extension, those previously treated with Hydrochlorothiazide (HCTZ) 12.5 or 25 mg in addition to aliskiren 300 mg/valsartan 320 mg were treated with aliskiren 300 mg/valsartan 320 mg/HCTZ 25 mg in the extension. Those patients who had not received HCTZ during the core study were treated with aliskiren 300 mg/valsartan 320 mg/HCTZ 12.5 mg.
  The HCTZ 12.5 mg dose could be increased to HCTZ 25 mg if the mean sitting Systolic Blood Pressure (msSBP) was ≥140 mmHg and/or the mean sitting Diastolic Blood Pressure (msDBP) was ≥90 mmHg for 2 consecutive visits.
  Interventions: Drug: Aliskiren; Drug: Valsartan; Drug: Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg
Drug: Valsartan — Valsartan 320 mg
Drug: Hydrochlorothiazide (HCTZ) — Hydrochlorothiazide (HCTZ) 12.5-25 mg
  Arms: Extension Treatment

SUMMARY:
Assessment of the long-term safety and tolerability of the combination of aliskiren and valsartan (300 mg/ 320 mg) in patients with high blood pressure,followed by assessment of long-term safety and tolerability of the combination of aliskiren/valsartan/Hydrochlorothiazide(HCTZ).

ELIGIBILITY:
Inclusion Criteria: -

* Male and female outpatients 18 years of age and older.
* For newly diagnosed/untreated patients with essential hypertension defined as msDBP ≥ 90 and < 110 mmHg at Visit 1 and Visit 4
* For previously treated patients with essential hypertension defined as msDBP ≥ 90 and < 110 mmHg after 2 to 4 weeks of washout (Visit 4)
* Patients who were eligible and able to participate in the study and who consented to do so after the purpose and nature of the investigation had been clearly explained to them (written informed consent).

Exclusion Criteria:

* Severe hypertension (msDBP ≥ 110 mmHg and/or msSBP ≥ 180 mmHg)
* Women of child-bearing potential, unless they met definition of post-menopausal or were using acceptable methods of contraception.
* History or evidence of a secondary form of hypertension.
* History of hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Investigative Centers, San Diego, California, United States
- Investigative Centers, Canada, Canada
- Investigative Centers, Germany, Germany
- Investigative Centers, Netherlands, Netherlands

REFERENCES:
- [Derived] Chrysant SG, Murray AV, Hoppe UC, Dattani D, Patel S, Ritter S, Zhang J. Long-term safety and efficacy of aliskiren and valsartan combination with or without the addition of HCT in patients with hypertension. Curr Med Res Opin. 2010 Dec;26(12):2841-9. doi: 10.1185/03007995.2010.528282. Epub 2010 Nov 9. PMID 21062137

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Treatment: Oral pills of aliskiren 150 mg /valsartan 160 mg in combination for 2-weeks. The aliskiren 300 mg /valsartan 320 mg in combiniation for 52-weeks, optional addition of HCTZ 12.5 mg starting from Week 10 if the blood pressure was uncontrolled (msSBP ≥ 140 and/or msDBP ≥ 90 mmHg). The dose of HCTZ 12.5 mg could be increased to 25 mg if blood pressure remained uncontrolled.
- Extension Treatment: For patients entering into extension, those previously treated with HCTZ (12.5 or 25 mg) in addition to aliskiren 300 mg/valsartan 320 mg were treated with aliskiren 300 mg/valsartan 320 mg/HCTZ 25 mg in the extension.
  Those patients who had not received HCTZ during the core study were treated with aliskiren 300 mg/valsartan 320 mg/HCTZ 12.5 mg.
  The HCTZ 12.5 mg dose could be increased to HCTZ 25 mg if the msSBP was ≥140 mmHg and/or the msDBP was ≥90 mmHg for 2 consecutive visits.
Period: Core
Arm/Group | Core Treatment | Extension Treatment
Started | 601 | 0
Completed | 486 | 0
Not Completed | 115 | 0
Not completed — Adverse Event | 40 | 0
Not completed — Abnormal laboratory value(s) | 3 | 0
Not completed — Unsatisfactory therapeutic effect | 23 | 0
Not completed — Condition no longer requires study drug | 4 | 0
Not completed — Patient withdrew consent | 15 | 0
Not completed — Lost to Follow-up | 23 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Protocol Deviation | 6 | 0
Period: Extension
Arm/Group | Core Treatment | Extension Treatment
Started | 0 | 162
Completed | 0 | 145
Not Completed | 0 | 17
Not completed — Adverse Event | 0 | 6
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Patient withdrew consent | 0 | 5
Not completed — Unsatisfactory therapeutic effect | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Core Treatment
Number analyzed (Participants) | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271
  Male | 330

OUTCOME MEASURES:

1. Primary Outcome: Overall Percentage of Patients With Adverse Events
Time Frame: Month 12
Population: Treated population: All patients who received at least one dose of Aliskiren/Valsartan
Measure: Number; unit: percentage of patients
Groups:
- Core Treatment- Aliskiren/Valsartan & Aliskiren/Valsartan/HCTZ: Oral pills of aliskiren 150 mg /valsartan 160 mg in combination for 2-weeks. The aliskiren 300 mg /valsartan 320 mg in combiniation for 52-weeks, optional addition of HCTZ 12.5 mg starting from Week 10 if the blood pressure was uncontrolled (msSBP ≥ 140 and/or msDBP ≥ 90 mmHg). The dose of HCTZ 12.5 mg could be increased to 25 mg if blood pressure remained uncontrolled.
Arm/Group | Core Treatment- Aliskiren/Valsartan & Aliskiren/Valsartan/HCTZ
Number analyzed (Participants) | 601
percentage of patients | 76.2

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure.
Time Frame: Baseline and Weeks 2, 4, 6, 10, 14, 18, 28, 41, and 54
Population: Treated population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Core Treatment
Number analyzed (Participants) | 601
mmHg
  Week 2 (Visit 5) | -7.9 (7.14)
  Week 4 (Visit 6) | -10.8 (7.83)
  Week 6 (Visit 7) | -11.8 (8.09)
  Week 10 (Visit 8) | -12.5 (8.26)
  Week 14 (Visit 9) | -13.7 (7.87)
  Week 18 (Visit 10) | -15.0 (8.00)
  Week 28 (Visit 11) | -15.2 (7.24)
  Week 41 (Visit 12) | -15.2 (7.60)
  Week 54 (Visit 13) | -14.2 (7.96)
  Endpoint (value at week 54 or LOCF) | -13.4 (8.75)

3. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure.
Time Frame: Baseline and Weeks 2, 4, 6, 10, 14, 18, 28, 41 and 54
Population: Treated population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Core Treatment
Number analyzed (Participants) | 601
mmHg
  Week 2 (Visit 5) | -11.0 (12.42)
  Week 4 (Visit 6) | -15.0 (14.03)
  Week 6 (Visit 7) | -17.6 (14.10)
  Week 10 (Visit 8) | -18.4 (14.37)
  Week 14 (Visit 9) | -20.7 (13.42)
  Week 18 (Visit 10) | -22.6 (14.01)
  Week 28 (Visit 11) | -24.3 (13.70)
  Week 41 (Visit 12) | -24.3 (13.27)
  Week 54 (Visit 13) | -22.3 (14.51)
  Endpoint (value at week 54 or LOCF) | -20.5 (16.40)

4. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control Target of < 140/90 mmHg
Time Frame: .Weeks 2, 4, 6, 10, 14, 18, 28, 41, and 54
Population: Treated population
Measure: Number; unit: Percentage of patients
Arm/Group | Core Treatment
Number analyzed (Participants) | 601
Percentage of patients
  Week 2 (Visit 5) | 32.8
  Week 4 (Visit 6) | 45.9
  Week 6 (Visit 7) | 52.4
  Week 10 (Visit 8) | 60.8
  Week 14 (Visit 9) | 68.7
  Week 18 (Visit 10) | 76.4
  Week 28 (Visit 11) | 77.9
  Week 41 (Visit 12) | 78.2
  Week 54 (Visit 13) | 71.7
  Endpoint (value at week 54 or LOCF) | 66.9

5. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure
Time Frame: Baseline and Month 18
Population: Treated population
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Extension Treatment: All patients receiving aliskiren / valsartan / HCTZ in extension study.
Arm/Group | Extension Treatment
Number analyzed (Participants) | 179
mmHg | -18.3 (8.52)

6. Primary Outcome: Overall Percentage of Patients With Adverse Events
Description: adverse event data obtained from both the core study and the 6 month extension study.
Time Frame: Month 18
Measure: Number; unit: percentage of patients
Groups:
- Core and Extension Treatment - Aliskiren/Valsartan/HCTZ: All patients receiving aliskiren / valsartan / HCTZ during either core or extension study.
Arm/Group | Core and Extension Treatment - Aliskiren/Valsartan/HCTZ
Number analyzed (Participants) | 310
percentage of patients | 61.6

7. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure
Time Frame: Baseline and Month 18
Population: Treated population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Extension Treatment
Number analyzed (Participants) | 179
mmHg | -28.8 (14.80)

8. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control Target of < 140/90 mmHg in Extension Treatment
Time Frame: Month 18
Population: Treated population
Measure: Number; unit: Percentage of patients
Arm/Group | Extension Treatment
Number analyzed (Participants) | 179
Percentage of patients | 86.6

ADVERSE EVENTS:
Time Frame: 18 months
Description: All patients who received at least one dose of study medication.
Groups:
- Core Period: Aliskiren 150 mg / Valsartan 160 mg Alone: Core Period: Aliskiren 150 mg /Valsartan 160 mg alone
- Core Period: Aliskiren 300 mg / Valsartan 320 mg Alone: Core Period: Aliskiren 300 mg /Valsartan 320 mg alone
- Core Period: Aliskiren / Valsartan: Core Period: Aliskiren/Valsartan
- Core and Extension: Aliskiren / Valsartan / HCTZ 12.5 mg: Core and Extension: Aliskiren / Valsartan / HCTZ 12.5 mg
- Core and Extension: Aliskiren / Valsartan / HCTZ 25 mg: Core and Extension: Aliskiren/Valsartan/HCTZ 25 mg
- Core and Extension: Total: Core and Extension: Total includes all study patients, treated with Aliskiren/Valsartan or Aliskiren//valsartan/HCTZ during core or extension.
Arm/Group | Core Period: Aliskiren 150 mg / Valsartan 160 mg Alone | Core Period: Aliskiren 300 mg / Valsartan 320 mg Alone | Core Period: Aliskiren / Valsartan | Core and Extension: Aliskiren / Valsartan / HCTZ 12.5 mg | Core and Extension: Aliskiren / Valsartan / HCTZ 25 mg | Core and Extension: Total
Serious Adverse Events (participants affected / at risk) | 3/601 | 14/585 | 17/601 | 3/306 | 6/137 | 26/601
Other Adverse Events (participants affected / at risk) | 49/601 | 185/585 | 215/601 | 47/306 | 26/137 | 251/601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Period: Aliskiren 150 mg / Valsartan 160 mg Alone (N=601) | Core Period: Aliskiren 300 mg / Valsartan 320 mg Alone (N=585) | Core Period: Aliskiren / Valsartan (N=601) | Core and Extension: Aliskiren / Valsartan / HCTZ 12.5 mg (N=306) | Core and Extension: Aliskiren / Valsartan / HCTZ 25 mg (N=137) | Core and Extension: Total (N=601)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Period: Aliskiren 150 mg / Valsartan 160 mg Alone (N=601) | Core Period: Aliskiren 300 mg / Valsartan 320 mg Alone (N=585) | Core Period: Aliskiren / Valsartan (N=601) | Core and Extension: Aliskiren / Valsartan / HCTZ 12.5 mg (N=306) | Core and Extension: Aliskiren / Valsartan / HCTZ 25 mg (N=137) | Core and Extension: Total (N=601)
Diarrhoea (Gastrointestinal disorders) | 8 | 27 | 34 | 9 | 1 | 42
Bronchitis (Infections and infestations) | 3 | 24 | 27 | 6 | 3 | 34
Nasopharyngitis (Infections and infestations) | 6 | 39 | 43 | 10 | 6 | 54
Upper respiratory tract infection (Infections and infestations) | 2 | 25 | 28 | 9 | 2 | 38
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 19 | 21 | 5 | 6 | 32
Dizziness (Nervous system disorders) | 15 | 39 | 49 | 6 | 7 | 61
Headache (Nervous system disorders) | 16 | 33 | 45 | 4 | 2 | 50
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 23 | 24 | 5 | 5 | 31

LIMITATIONS AND CAVEATS:
Open label study with no comparator treatment/arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.